CLINICAL TRIAL: NCT01650168
Title: Prospective Controlled Cohort Study on the Safety of a Monophasic Oral Contraceptive Containing Nomegestrol Acetate (2.5mg) and 17ß-estradiol (1.5mg)
Acronym: PRO-E2
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Theramex (Industry)
Responsible Party: Sponsor
Other Study IDs: ZEG2013_08
Record Dates: First submitted 2012-07-13; First posted 2012-07-26 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Contraception
Keywords: NOMAC-E2; Nomegestrol acetate; Estradiol; Levonorgestrel; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NOMAC-E2: New users of NOMAC-E2
- LNG-COCs: New users of levonorgestrel-containing COCs

SUMMARY:
This study compares the risks of short- and long-term use of NOMAC-E2 (containing a fixed dose of nomegestrol acetate and estradiol) compared with levonorgestrel-containing combined oral contraceptives (COC-LNG) in a study population representative of the actual users of the individual preparations.

DETAILED DESCRIPTION:
NOMAC-E2 is a novel monophasic oral contraceptive containing a fixed dose of nomegestrol acetate (2.5mg) and 17ß-estradiol (1.5mg) which is taken for 24 days followed by 4 days of placebo. The most relevant adverse clinical outcome that has been linked to the use of COCs is venous thromboembolism (VTE). Data from randomized clinical trials did not show any serious health concerns for NOMAC-E2. However, the statistical power to detect rare adverse events is limited in these studies.

PRO-E2 is a large, prospective, controlled, long-term active surveillance study to investigate the safety of NOMAC-E2 with regard to the outcomes of interest. This study follows the European Active Surveillance (EURAS) design methodology with some modifications due to country- and product-specific characteristics. The outcomes of interest will be validated via the attending physicians. A multi-faceted follow-up procedure will ensure a low loss to follow-up rate. This study will involve women from Europe and Australia who will be followed for up to 2 years. Data analysis will include multivariable techniques such as Cox regression.

ELIGIBILITY:
Inclusion Criteria:

* First ever user of a COC ("starter")
* User who restarts hormonal contraceptive use with a COC (same COC as before or a new COC) after an intake break of at least two months ("restarters")
* Women willing to participate in the active surveillance

Exclusion Criteria:

- Women who do not understand the major aspects of the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women using oral contraceptives
Sampling Method: Non-Probability Sample
Enrollment: 101498 (Actual)
Dates: Start 2012-07; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolisms (VTE) | Within 2 years

SECONDARY OUTCOMES:
Arterial thromboembolisms (ATE) | Within 2 years
Depressive disorders | Within 2 years
Cholelithiasis | Within 2 years
Inflammatory bowel disease | Within 2 years
Short- and long-term fertility | Within 2 years
Drug utilization pattern | Within 2 years
Pregnancy outcomes | Within 2 years
Weight change | Within 2 years
General hepatobiliary disorders | Within 2 years
Acne | Within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research, Berlin, Germany
Locations (1):
- Center for Epidemiology and Health Research Berlin, Berlin, Germany